CLINICAL TRIAL: NCT01549379
Title: Dynamic Contrast Enhanced Computed Tomography (DCE-CT) to Assess Lymph Node Metastases in Head and Neck Cancer: A Prospective Study
Brief Title: Dynamic Contrast Enhanced Computed Tomography (CT) for Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Regional Cancer Program, Canada (Other)
Responsible Party: Principal Investigator, David Palma, Radiation Oncologist/Clinician Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UWO18826; 18826 (Other: REB)
Record Dates: First submitted 2012-02-24; First posted 2012-03-09 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; Radiation; Chemotherapy; Surgery; Dynamic contrast enhanced computed tomography
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical patients (Active Comparator): This group will consist of 15 patients with locally advanced HNSCC of the oral cavity, larynx or hypopharynx presenting with adenopathy ≥ 1 cm where the recommended treatment is surgical resection of the primary malignancy with bilateral neck dissection. These patients will receive a DCE-CT scan of the head and neck prior to surgery.
  Interventions: Radiation: Dynamic Contrast Enhanced CT scan
- Chemoradiation Patients (Active Comparator): This group will consist of 15 patients with locally advanced HNSCC with lymph nodes ≥3 cm in which chemoradiotherapy is the primary treatment as per standard of care. This group will be composed of patients with a primary malignancy originating in the nasopharynx, oropharynx, hypopharynx or larynx. Pre-treatment DCE-CT of neck will be obtained. The standard therapy, radiation and chemotherapy, will be administered and the patients will have standard follow up. A post-treatment DCE-CT of neck will be obtained 8-10 weeks after treatment along with standard CT neck.
  Interventions: Radiation: Dynamic Contrast Enhanced CT scan

INTERVENTIONS:
Radiation: Dynamic Contrast Enhanced CT scan — The neck will be scanned using 120 kVp, 50 mAs, 8 x 5 mm slices at intervals of 2.8 - 3.0 s for 3 min. Contrast (e.g. Visipaque 320) at a dosage of 0.7 ml/kg is injected at 4 ml/s through an antecubital vein after a delay of 6 s from start of scanning.

SUMMARY:
For patients undergoing treatment for head and neck cancer, this study will use dynamic contrast-enhanced CT scans to try to determine which lymph nodes in the neck contain cancer and require surgical removal.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide informed consent
* ECOG performance status 0-2
* Histologically confirmed squamous cell carcinoma (includes variants such as verrucous carcinoma, spindle cell carcinoma, carcinoma NOS) of the head and neck
* Tumor stage: Any (T1-T4)
* Nodal stage:

  * N2 or N3 (≥ 3 cm) on pre-treatment imaging for radiotherapy cohort (higher likelihood of requiring neck dissection);
  * N1-N3 for surgery cohort. N0 admissible for T4 tumors.
* Patient assessed at head and neck multidisciplinary clinic (with assessment by radiation oncologist and surgeon), with recommendation for definitive chemoradiation therapy (n=15) or surgery (n=15)

Exclusion Criteria:

* Prior history of head and neck cancer within 5 years
* Prior head and neck radiation at any time
* Metastatic disease, or imaging findings suspicious for metastases
* Prior invasive malignant disease unless disease-free for at least 5 years or more, with the exception of non-melanoma skin cancer.
* Pregnant or lactating women
* Contraindication to DCE-CT (e.g. contrast allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of DCE-CT in predicting the presence of residual lymph node disease after the completion of chemotherapy | 8-10 weeks post treatment

SECONDARY OUTCOMES:
Sensitivity and specificity of DCE-CT in predicting presence of lymph node disease at surgery | Approximately 2-6 weeks after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: David A Palma, MD, MSc, PhD, Principal Investigator — London Regional Cancer Program
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada